CLINICAL TRIAL: NCT02470858
Title: Effect of Triple Direct Acting Antiviral Agents (DAAs) for Non-cirrhotic Subjects With Chronic HCV G1b Infection
Brief Title: Triple DAAs Regimen in Treating Non-cirrhotic HCV GT1b Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&H_Triple Therapy_1
Record Dates: First submitted 2015-06-05; First posted 2015-06-12 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — Sofosbuvir; ledipasvir; ledipasvir, sofosbuvir drug combination; asunaprevir; daclatasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LDV/SOF+ASV (Experimental): Participants with genotype 1b HCV infection will receive LDV/SOF FDC + ASV 3 weeks.
  Interventions: Drug: LDV/SOF+ASV
- SOF+DCV+SMV (Experimental): Participants with genotype 1b HCV infection will receive SOF + DCV + SMV for 3 weeks.
  Interventions: Drug: SOF+DCV+SMV
- SOF+DCV+ASV (Experimental): Participants with genotype 1b HCV infection will receive SOF + DCV + ASV for 3 weeks
  Interventions: Drug: SOF+DCV+ASV

INTERVENTIONS:
Drug: LDV/SOF+ASV — Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed-dose combination (FDC) tablet; administered orally once daily; Asunaprevir (ASV) 200mg, administered orally twice daily.
  Other Names: GS-7977; PSI-7977; GS-5885; Harvoni®; BMS-650032; Sunvepra®
  Arms: LDV/SOF+ASV
Drug: SOF+DCV+SMV — Sofosbuvir (SOF) 400 mg tablet administered orally once daily; Daclatasvir (DCV) 60 mg tablet administered orally once daily; Simeprevir (SMV) 150 mg tablet orally once daily.
  Other Names: GS-7977; PSI-7977; Sovaldi®; BMS-790052; Daklinza®; TMC435; OLYSIO®
  Arms: SOF+DCV+SMV
Drug: SOF+DCV+ASV — Sofosbuvir (SOF) 400 mg tablet administered orally once daily; Daclatasvir (DCV) 60 mg tablet administered orally once daily; Asunaprevir (ASV) 200mg, administered orally twice daily.
  Other Names: GS-7977; PSI-7977; Sovaldi®; BMS-790052; Daklinza®; BMS-650032; Sunvepra®
  Arms: SOF+DCV+ASV

SUMMARY:
The study is designed to test the hypothesis that the addition of a protease inhibitor to dual NS5a-NS5B nucleoside prodrug analog will enhance antiviral efficacy and hence shorten the treatment duration to 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years, with chronic genotype 1b HCV infection;
* HCV RNA level > 10,000 and < 10,000,000 IU/ml at Screening;
* Rapid response to triple DAAs therapy with less than 500 IU/ml plasma HCV RNA level at Day 2;
* No evidence of cirrhosis. Cirrhosis defined as any 1 of the following, within 6 months of study entry:

  1. Liver biopsy showing cirrhosis;
  2. Fibroscan showing cirrhosis or results>12.5 kPa ;
  3. FibroTest® score >0.75 and an aspartate aminotransferase (AST): platelet ratio index (APRI) >2 during screening.

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner;
* HIV or chronic hepatitis B virus (HBV) infection;
* Hematologic or biochemical parameters at Screening outside the protocol-specified requirements;
* Active or recent history (≤ 1 year) of drug or alcohol abuse;
* Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers);
* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained virologic response 12 weeks after discontinuation of therapy (SVR12) | Post treatment Week 12
  SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after last dose of study drug.
Proportion of participants with adverse events leading to permanent discontinuation of study drug(s) | Baseline up to Week 24

SECONDARY OUTCOMES:
Proportion of participants with unquantifiable HCV viral load at specified time points during and after treatment. | Baseline up to Week 24
HCV RNA levels and change during and after treatment. | Baseline up to Week 24
Proportion of participants with on-treatment virologic breakthrough and relapse | Baseline up to Week 24
  Viral breakthrough is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) during treatment, but did not achieve a sustained virologic response (SVR). Viral relapse is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) within 4 weeks of end of treatment, but did not achieve an SVR.

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, Principal Investigator — Humanity and Health GI and Liver Centre
Locations (1):
- Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Lau G, Benhamou Y, Chen G, Li J, Shao Q, Ji D, Li F, Li B, Liu J, Hou J, Sun J, Wang C, Chen J, Wu V, Wong A, Wong CL, Tsang ST, Wang Y, Bassit L, Tao S, Jiang Y, Hsiao HM, Ke R, Perelson AS, Schinazi RF. Efficacy and safety of 3-week response-guided triple direct-acting antiviral therapy for chronic hepatitis C infection: a phase 2, open-label, proof-of-concept study. Lancet Gastroenterol Hepatol. 2016 Oct;1(2):97-104. doi: 10.1016/S2468-1253(16)30015-2. Epub 2016 Jul 25. PMID 27917405